CLINICAL TRIAL: NCT05469815
Title: Lost Children Society (LCS), Metacognitive Training Integrated Into an Online Therapeutic Tabletop Role-playing Game for Early-onset Schizophrenia Patients : a Pilot Study on Feasibility
Brief Title: Lost Children Society (LCS), Online Therapeutic Tabletop Role-playing Game for Early-onset Schizophrenia Patients
Acronym: TTRPG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: * The tool's target population has changed.
  * It proved impossible to recruit 16 individuals from the original target population, despite the initial commitment of expert centres.
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHD22_0001
Record Dates: First submitted 2022-06-23; First posted 2022-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Metacognitive Training; Early-onset Schizophrenia; Therapeutic TableTop Role Playing Game; Psychoeducational program; Lost Children Society
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lost Children Society Game (Experimental): Online therapeutic role-playing session
  Interventions: Behavioral: Lost Children Society Game

INTERVENTIONS:
Behavioral: Lost Children Society Game — 36 online therapeutic role-playing sessions spread over 36 weeks, one session per week

SUMMARY:
The Lost Children Society (LCS) is a Therapeutic TableTop Role-Playing Game specifically developed for early-onset schizophrenia patient.

It is performed online via a secure teleconsultation and videoconference platform.

Patients are connected from their home, on their personal computer or tablet, equipped with headsets with microphone.

This study aims to validate the feasibility of this online Therapeutic TableTop Role Playing Game.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early onset schizophrenia
* Patient who has the capacity to understand the protocol and to perform evaluations
* Written informed consent to participate in the study given by the patient or by the parental authority of the minor patient.
* Patient with social security coverage

Exclusion Criteria:

* Intelligence quotient<70 on Wechsler Adults Intelligence Scale-IV (for 17+ years) or the Wechsler Intelligence Scale for Children V (for 15-16 years).
* Personal history of head trauma, neurological disorder, genetic disease.
* Co-morbidities: major depressive episode or post-traumatic stress disorder unresolved or resolved within the last 6 months.
* Lack of mastery or access to a computer or personal tablet in autonomy
* Therapeutic history of metacognitive training.
* Patient under guardianship, curators or legal protection
* Patient going through a period of exacerbation of positive or negative psychotic signs likely to lead to a full-time hospitalization in a specialized environment within the next 3 months

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Overall feasibility of the Game | 10 month
  Effective participation of the patient - feasibility will be defined by the number of effective sessions > or = 29

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan PIONNIER, Principal Investigator — EPSM de Vendée Georges Mazurelle

IPD SHARING:
Plan to Share IPD: No